CLINICAL TRIAL: NCT05929105
Title: Short-term Outcome of Artificial Intelligence-assisted Preoperative Three-dimensional Planning of Total Hip Arthroplasty for Developmental Dysplasia of the Hip Compared With Traditional Surgery
Brief Title: AI-assisted Preoperative Planning Technology for THA for DDH
Status: Completed | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Principal Investigator, Peng Li, Deputy Director, General Hospital of Ningxia Medical University
Other Study IDs: lipeng2023
Record Dates: First submitted 2023-06-05; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group
  Interventions: Procedure: artificial intelligence (AI)-assisted three-dimensional preoperative planning technology
- control group
  Interventions: Other: X-ray film template for 2D planning

INTERVENTIONS:
Procedure: artificial intelligence (AI)-assisted three-dimensional preoperative planning technology — In the AI planning group, AI was used to assist in the 3D planning to complete the preoperative design. Preoperative planning was performed by two experienced surgeons and without the chief physician to ensure that the results of the preoperative planning did not affect the selection of intraoperative procedures and prosthesis size.
  Groups: observation group
Other: X-ray film template for 2D planning — A traditional X-ray film template was used to complete the preoperative design in the traditional planning group. The position and size of the prosthesis, the level of femoral neck osteotomy, the length of the LLs and the restoration of eccentricity were estimated by X-ray. A plastic template provided by the manufacturer was used to take the line of the lower edge of the teardrop on both sides as the horizontal reference line, and the acetabular template was placed at 40 abduction on the inner edge of the teardrop so that the lower edge of the acetabular cup was adjacent to the teardrop. An appropriate type of acetabular component was selected to fill the acetabulum and maintain coverage, and the femoral component that best matched the femoral medullary cavity was chosen. The height of the osteotomy was determined, and the planning model was recorded after the surgeons were happy with the placement and outcome.
  Groups: control group

SUMMARY:
In this study, the investigators retrospectively collected DDH case data of THA assisted by AI 3D planning and THA assisted by traditional planning. The compliance between preoperative planning and the type of prosthesis used in the operation, the position of the acetabular prosthesis, the correction of LLD and the postoperative joint function score were analysed to evaluate the short-term effect of AI combined with preoperative 3D planning in THA for DDH.

ELIGIBILITY:
Inclusion Criteria:

* DDH was diagnosed by clinical signs and imaging examination, and a primary THA was planned;
* the patient had persistent unilateral hip pain, which seriously affected their quality of life;
* the standard posterolateral approach was used;
* the contralateral hip was normal or had received THA;
* the proximal femoral Dorr classification was type A or B;
* The acetabular classification was Crowe type Ⅰ, Ⅱ, Ⅲ or IV;
* all patients were treated with the bioartificial hip joint PINNACLE® cup or SUMMIT® stem, developed by Johnson & Johnson Biological.

Exclusion Criteria:

* preoperative and postoperative imaging examinations did not meet the evaluation criteria (non-standard double-hip anteroposterior film, acetabular angle and LL length could not be accurately measured);
* severe osteoporosis, tumour or metabolic disease around the affected hip joint;
* spinal deformity by other causes or a history of lumbar internal fixation;
* external deformity of the affected hip joint in the lower extremity;
* neuromuscular insufficiency (with hip abduction weakness and poliomyelitis);
* severe disease with intolerance to surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with DDH who underwent unilateral primary THA between January 2020 and July 2022 in the orthopaedic department.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Type of acetabular cup and femoral stem | 31 months
  Accuracy analysis of planning model and the practical model
Difference in the length of lower limbs before and after surgery | 31 months
  Prove the accuracy of the artificial intelligence planning group

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China